CLINICAL TRIAL: NCT06924047
Title: The Clinical Performance of Two Dentine Replacement Materials in Deep Occlusal Cavities: A Randomized Clinical Trial
Brief Title: The Clinical Performance of Two Dentine Replacement Materials in Deep Occlusal Cavities (Randomized)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dalia Sameh Fawzi (Other)
Responsible Party: Sponsor-Investigator, Dalia Sameh Fawzi, Principle Investigator, Future University in Egypt
Organization: Future University in Egypt (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Restoring Deep Occlusal Cavity
Record Dates: First submitted 2025-03-18; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Class I Cavities in High Caries Risk; Class I Composite Restorations; Randomized Clinical Trial; Occlusal Caries; Fiber Reinforced Composite; Injectable Composite; Composite Restoration; Composite Resins
Keywords: occlusal caries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bioactive injectable composite (Active Comparator): bioactive injectable composite placed as a dentine substitute
  Interventions: Other: Beautifil Flow Plus X
- Short fiber reinforced composite (Active Comparator): Short fiber reinforced composite added as a dentine substitute
  Interventions: Other: EverX Flow

INTERVENTIONS:
Other: Beautifil Flow Plus X — Shofu's Beautifil Flow Plus X F00 a advanced bioactive injectable composite
  Arms: Bioactive injectable composite
Other: EverX Flow — Short fiber reinforced composite
  Arms: Short fiber reinforced composite

SUMMARY:
Higher mechanical properties are needed to restore structurally compromised posterior teeth, short fiber reinforced resin composite and injectable bioactive resin composites provide superior properties to flowable composites that were traditionally used to improve adaptation in deep cavities below the packable resin composite restorations. Thus, this study was designed to assess the clinical outcome of high strength dentine substitute materials.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients aged (20-50)
2. Medically free
3. Good oral hygiene (Plaque index ≤2 (Moderate accumulation with plaque in the sulcus))
4. Patients accepting to participate in the study.
5. Teeth of normal appearance and morphology
6. Maxillary and mandibular molar teeth with deep class Ⅰ carious lesions extending into the inner third of dentin.

Exclusion Criteria:

1. Patients <20 and >50.
2. Teeth with proximal lesions.
3. Patients with bad oral hygiene (Plaque index >2).
4. Systematic disease that may interfere with the study.
5. Patients with xerostomia.
6. Presence of any abnormal occlusal habits (bruxism, nail biting, clenching).
7. Patients undergoing or will start orthodontic treatment.
8. Pregnancy.
9. Teeth with signs or symptoms of irreversible pulpitis.
10. Non-vital, fractured or cracked teeth.
11. Teeth with secondary caries.
12. Periodontally compromised teeth.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Fracture | T1: 1 week T2: 6months T3: 12 months
  1. Clinically excellent/very good (sufficient): Restoration is completely present without deficiencies detectable after air drying.
  2. Clinically good (sufficient): Restoration is completely present with minor deficiencies detectable after air drying
  3. Clinically satisfactory (sufficient): Restoration is present with deficiencies detectable without air drying
  4. Clinically unsatisfactory (partially insufficient): Localized but severe deficiencies regarding fracture and retention
  5. Clinically poor (entirely insufficient): Generalized severe deficiencies

SECONDARY OUTCOMES:
Recurrent caries | T1: 1 week T2: 6months T3: 12 months
  1. Clinically excellent/very good (sufficient): No caries/demineralization at the restoration margin detectable after air drying.
  2. Clinically good (sufficient): First visible signs of a non-cavitated caries lesion at the restoration margin detectable after air drying.
  3. Clinically satisfactory (sufficient): Established, non- cavitated caries lesion or microcavity at the restoration margin detectable without air drying.
  4. Clinically unsatisfactory (partially insufficient):
     Localized dentin cavity at the restoration margin.
  5. Clinically poor (entirely insufficient): Extensive dentin cavity at the restoration margin.
Post operative sensitivity | T1: 1 week T2: 6months T3: 12 months
  1. Clinically excellent/very good (sufficient): No Postoperative hypersensitivity.
  2. Clinically good (sufficient): Minor postoperative hypersensitivity.
  3. Clinically satisfactory (sufficient) Distinct "moderate" postoperative hypersensitivity.
  4. Clinically unsatisfactory (partially insufficient): Severe "persistent" postoperative hypersensitivity.
  5. Clinically poor (entirely insufficient): Extreme postoperative hypersensitivity "Irreversible pulpitis".

REFERENCES:
- [Background] Yao Y, Luo A, Hao Y. Selective versus stepwise removal of deep carious lesions: A meta-analysis of randomized controlled trials. J Dent Sci. 2023 Jan;18(1):17-26. doi: 10.1016/j.jds.2022.07.021. Epub 2022 Aug 21. PMID 36643250
- [Background] Schwendicke F, Frencken JE, Bjorndal L, Maltz M, Manton DJ, Ricketts D, Van Landuyt K, Banerjee A, Campus G, Domejean S, Fontana M, Leal S, Lo E, Machiulskiene V, Schulte A, Splieth C, Zandona AF, Innes NP. Managing Carious Lesions: Consensus Recommendations on Carious Tissue Removal. Adv Dent Res. 2016 May;28(2):58-67. doi: 10.1177/0022034516639271. PMID 27099358
- [Background] Rusnac ME, Gasparik C, Irimie AI, Grecu AG, Mesaros AS, Dudea D. Giomers in dentistry - at the boundary between dental composites and glass-ionomers. Med Pharm Rep. 2019 Apr;92(2):123-128. doi: 10.15386/mpr-1169. Epub 2019 Apr 25. PMID 31086838
- [Background] Reis A, Carrilho M, Breschi L, Loguercio AD. Overview of clinical alternatives to minimize the degradation of the resin-dentin bonds. Oper Dent. 2013 Jul-Aug;38(4):E1-E25. doi: 10.2341/12-258-LIT. Epub 2013 Mar 25. PMID 23527523
- [Background] Qin D, Hua F, John MT. GLOSSARY FOR DENTAL PATIENT-CENTERED OUTCOMES. J Evid Based Dent Pract. 2024 Jan;24(1S):101951. doi: 10.1016/j.jebdp.2023.101951. Epub 2023 Nov 5. PMID 38401954
- [Background] Ozer F, Patel R, Yip J, Yakymiv O, Saleh N, Blatz MB. Five-year clinical performance of two fluoride-releasing giomer resin materials in occlusal restorations. J Esthet Restor Dent. 2022 Dec;34(8):1213-1220. doi: 10.1111/jerd.12948. Epub 2022 Aug 7. PMID 35934807
- [Background] Maillet C, Decup F, Dantony E, Iwaz J, Chevalier C, Gueyffier F, Maucort-Boulch D, Grosgogeat B, Le Clerc J. Selected and simplified FDI criteria for assessment of restorations. J Dent. 2022 Jul;122:104109. doi: 10.1016/j.jdent.2022.104109. Epub 2022 Mar 26. PMID 35346772
- [Background] Ikeda I, Otsuki M, Sadr A, Nomura T, Kishikawa R, Tagami J. Effect of filler content of flowable composites on resin-cavity interface. Dent Mater J. 2009 Nov;28(6):679-85. doi: 10.4012/dmj.28.679. PMID 20019418
- [Background] Hoefler V, Nagaoka H, Miller CS. Long-term survival and vitality outcomes of permanent teeth following deep caries treatment with step-wise and partial-caries-removal: A Systematic Review. J Dent. 2016 Nov;54:25-32. doi: 10.1016/j.jdent.2016.09.009. Epub 2016 Sep 21. PMID 27664467
- [Background] Elderiny HM, Khallaf YS, Akah MM, Hassanein OE. Clinical Evaluation of Bioactive Injectable Resin Composite vs Conventional Nanohybrid Composite in Posterior Restorations: An 18-Month Randomized Controlled Clinical Trial. J Contemp Dent Pract. 2024 Aug 1;25(8):794-802. doi: 10.5005/jp-journals-10024-3737. PMID 39653674
- [Background] ElAziz RHA, ElAziz SAA, ElAziz PMA, Frater M, Vallittu PK, Lassila L, Garoushi S. Clinical evaluation of posterior flowable short fiber-reinforced composite restorations without proximal surface coverage. Odontology. 2024 Oct;112(4):1274-1283. doi: 10.1007/s10266-024-00905-5. Epub 2024 Feb 23. PMID 38393515
- [Background] European Society of Endodontology (ESE) developed by:; Duncan HF, Galler KM, Tomson PL, Simon S, El-Karim I, Kundzina R, Krastl G, Dammaschke T, Fransson H, Markvart M, Zehnder M, Bjorndal L. European Society of Endodontology position statement: Management of deep caries and the exposed pulp. Int Endod J. 2019 Jul;52(7):923-934. doi: 10.1111/iej.13080. PMID 30664240
- [Background] Bijelic-Donova J, Myyrylainen T, Karsila V, Vallittu PK, Tanner J. Direct Short-Fiber Reinforced Composite Resin Restorations and Glass-Ceramic Endocrowns in Endodontically Treated Molars: A 4 -Year Clinical Study. Eur J Prosthodont Restor Dent. 2022 Nov 30;30(4):284-295. doi: 10.1922/EJPRD_2333Bijelic-Donova12. PMID 35438265
- [Background] Battancs E, Sary T, Molnar J, Braunitzer G, Skolnikovics M, Schindler A, Szabo P B, Garoushi S, Frater M. Fracture Resistance and Microleakage around Direct Restorations in High C-Factor Cavities. Polymers (Basel). 2022 Aug 25;14(17):3463. doi: 10.3390/polym14173463. PMID 36080538